CLINICAL TRIAL: NCT01338805
Title: A Multicenter, Open-label, Follow-up Study to Evaluate the Long-term Safety and Tolerability of BGG492 TID as Adjunctive Therapy in Patients With Partial Onset Seizures Completing Double-blind, Placebo-controlled Study CBGG492A2207 or CBGG492A2211
Brief Title: Phase II BGG492 Capsule Extension for Partial Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBGG492A2212; 2010-021448-17 (EudraCT Number)
Record Dates: First submitted 2011-04-15; First posted 2011-04-20 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2016-03

CONDITIONS: Partial Onset Seizures
Keywords: Partial onset seizure; seizure frequency; nervous system diseases; central nervous system diseases; CNS; brain diseases; neurologic manifestations; adjunctive treatment; AEDs; antiepileptic drug
MeSH Terms: conditions — Nervous System Diseases; Central Nervous System Diseases; Brain Diseases; Neurologic Manifestations | interventions — selurampanel

ARMS (1):
- BGG492 (Experimental): hard gelatin capsule for oral administration at 50 mg TID, 100 mg TID or 150 mg TID
  Interventions: Drug: BGG492

INTERVENTIONS:
Drug: BGG492

SUMMARY:
This long-term extension study will assess the safety, tolerability and efficacy of BGG492 as adjunctive treatment in patients with partial onset seizures.

ELIGIBILITY:
Inclusion Criteria:

* Completed study CBGG492A2207, cooperated with the study procedures and did not experience persistent tolerability issues
* Outpatients ≥ 45 kg (99 lb) of weight
* Patient would like to continue BGG492 treatment and the investigator believes a reasonable benefit from the long-term administration of BGG492 may be expected
* Treated with a stable dose of one or a maximum of three licensed Antiepileptic drugs (AEDs)and are known to take their medication(s) as directed
* Will make themselves available for the study period and are able to record seizures and report adverse events themselves or have a caregiver who can record and report the events
* Provided written informed consent before any extension assessment is performed

Exclusion Criteria:

* Status epilepticus or seizure clusters occurring during study CBGG492A2207 or in the period between the end of study the double blind study and the start of study CBGG492A2212 for patients experiencing a treatment gap
* Have been treated with:
* Felbamate, unless treatment has been continuous for ≥ 2 years
* Vigabatrin during the 26 weeks prior to the first dose of open-label medication in the extension study
* Monoamine oxidase (MAO) inhibitors, tricyclic-antidepressants and narcotic analgesics
* L-Dopa formulations
* Use of concomitant medication that are potential inhibitors of Organic anion-transporting polypeptide (OATP) transporters
* No physical examination changes suggestive of progressive neurological changes during Study CBGG492A2207
* Used another investigational drug (other than BGG492) either at the time of enrollment in this extension study or within 5 half-lives prior to enrollment in this extension study
* History of hypersensitivity to the study drug or to drugs of similar chemical classes (e.g. sulfonamides) or had multiple drug allergies or one or more severe drug reactions to an Antiepileptic drugs (AEDs), including dermatological reactions
* Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the long-term safety and tolerability of BGG492 capsules during the maintenance period in patients suffering from partial onset seizures | 38 weeks
  By measuring the number and percent of patients having any AE (advent event) by primary system organ class and/or preferred term.
  By laboratory, vital sign, and ECG data, summary statistics of values and change from baseline

SECONDARY OUTCOMES:
To evaluate the efficacy over time by the change in partial seizure frequency original Baseline Period in the double-blind study CBGG492A2207 to the Open-label Extension Maintenance Phase. | 38 weeks
Responder rate: To evaluate the maintenance of efficacy by the change in responder rate and numbers of patients becoming seizure free from the original Baseline Period to the Open-label Extension Maintenance Phase. | 38 weeks
Seizure counts: To evaluate the maintenance of efficacy and safety as assessed in percent change of seizure frequency of BGG492 capsules from the original Baseline Period to the Open-label Extension Maintenance Phase. | 38 weeks
To evaluate long-term efficacy and safety by summarizing the number and percentage of patients who discontinue due to unsatisfactory therapeutic response effect and for all other reasons. | 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- United States (3):
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Hamilton, New Jersey
  - Novartis Investigative Site, Dallas, Texas
- Germany (5):
  - Novartis Investigative Site, Bernau
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Kehl-Kork
  - Novartis Investigative Site, Ulm
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kecskemét
  - Novartis Investigative Site, Szombathely
- Novartis Investigative Site, Warsaw, Poland
- Slovakia (2):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Košice
- Novartis Investigative Site, Seoul, Korea, South Korea

REFERENCES:
- See also: Results for CBGG492A2212 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=9223